CLINICAL TRIAL: NCT05172492
Title: Efficacy of Endocare Treatment at Home on Pain in Women With Chronic Pelvic-perineal Pain Related to Endometriosis. EndoHome.
Brief Title: Endocare for Pelvic-perineal Pain Related to Endometriosis Used at Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lucine (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-A02358-33
Record Dates: First submitted 2021-11-30; First posted 2021-12-29 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Endometriosis; Chronic Pain; Pelvic Pain
MeSH Terms: conditions — Endometriosis; Chronic Pain; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocare (Experimental)
  Interventions: Device: Endocare
- Digital control (Active Comparator)
  Interventions: Device: Digital control

INTERVENTIONS:
Device: Endocare — Endocare will be administred through a virtual reality headseat used one to twice a day.
  Arms: Endocare
Device: Digital control — Digital control will be administred through a virtual reality headseat used one to twice a day.
  Arms: Digital control

SUMMARY:
Women with endometriosis experience recurrent pelvic-perineal pain impairing the quality of life, among other things. Endometriosis-related pain negatively impacts the sexual, family and work life.

Apart from the usual painkillers, the doctor's current therapeutic arsenal is limited to hormonal contraceptives and surgery. As endometriosis-related treatments do not currently address all of the patients' problems, developing a new, effective, non-pharmaceutical treatment would make it possible to relieve the pain of these women.

Endocare treatment consists of visual and auditory therapeutic procedures for pelvic-perineal pain in patients with endometriosis.

Moreover, as Endocare is not a pharmacological molecule but a digital therapy, it would not increase the consumption of pharmacological agents. An analgesic effect of Endocare lasting several hours on chronic pelvic-perineal pain associated with endometriosis is expected.

The effects of the treatment will be compare to a digital control also integrated in a virtual reality headset identical to the one distributing Endocare allowing to maintain the blindness to the patients and the investigator on the treatment received.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age with diagnosed endometriosis (histology, imaging, clinical symptomatology) and/or adenomyosis.
* Women with at least 2 consecutive days per month of endometriosis-related pelvic-perineal pain of moderate to severe intensity (NS ≥ 4):

  * Women without amenorrhea: pain around the onset of menstruation.
  * Women with amenorrhea: most intense pain of the month.

Exclusion Criteria:

* Pregnant or nursing women.
* Women participating, or who have participated, in a clinical interventional study within 30 days prior to inclusion.
* Women with severe visual, auditory or cognitive impairment, color blindness, photosensitivity, epilepsy or motion sickness.
* Women whose pain is occasional and not present at each menstrual period.
* Women who have previously received virtual reality treatments.
* Women under judicial protection, guardianship, curatorship, protective mandate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Pain intensity change | Time points are before treatment (Time 0) and one hour after treatment (Time 1) during t five days (Day 1, Day 2, Day 3, Day 4, Day 5)
  The mean change in pain intensity assessed by a numeric rating scale (pain intensity numerical scale) between the pre-treatment measurement and one hour after the use of Endocare treatment, compared to the digital control during the five days of treatment.The pain scale is a 11-point numeric scale (0=no pain; 10=unbearable pain).

SECONDARY OUTCOMES:
Change in pain intensity | at wake-up and bedtime during the 5 days of treat (Day 1 to Day 5)
  Change in pain intensity assessed by numeric scale. The pain scale is a 11-point numeric scale (0=no pain; 10=unbearable pain).
Change in pain relief | At 1 hour (Time 1), 2 hours (Time 2) and 3 hours (Time 3) after treatment during the 5 days of treatment (Day 1 to Day 5)
  Change in pain relief assessed by Likert pain relief scale. Its a 5-point categorical scale (0: no relief, 1: slight relief, 2: moderate relief, 3: lots of relief and 4: complete relief)
Weighted average change in pain intensity | from pre-treatment (Time 0) to 2 hours (Time 2) and 3 hours (Time 3) post-treatment during the 5 days of treatment (Day 1 to Day 5)
  Weighted average change (based on number of treatments Endocare or control uses) in pain intensity assessed by numeric scale. The pain scale is a 11-point numeric scale (0=no pain; 10=unbearable pain).
Change in stress value | at wake-up and bedtime during the 5 days of treatment (Day 1 to Day 5)
  Change in stress assessed by Visual Analogue Scale (VAS). Visual Analogue Scale (VAS) consists of a small unmarked 100 mm ruler with ends labelled 'none' and 'as bad as possible'.
Change in fatigue value | at wake-up and bedtime during the 5 days of treatment (Day 1 to Day 5)
  Change in stress assessed by Visual Analogue Scale (VAS) and fatigue assessed by Pichot Scale. The Pichot scale evaluates 8 fatigue items ranging from 0 to 4 (0: not at all; 1: a little; 2: moderately; 3: a lot; 4: extremely)
Change in endometriosis-related quality of life | At inclusion visit Day 0 and at through study completion (Day 6), an average of one week
  Change in endometriosis-related quality of life assessed by Endometriosis Health Profile (EHP-5). The EHP-5 consists of 11 items ranging from "never" to "always"
Assessment of the predictive value of dramatization and catastrophizing thoughts | At the inclusion visit Day 0
  Assessment of the predictive value of dramatization and catastrophizing thoughts assessed by Patient catastrophizing scale (PCS) coonsisting of 13 items ranging from 0 to 4 (0= not at all; 1= to a slight degree; 2= to a moderate degree; 3= to a great degree; 4 = all the time).
Pain relief treatments | during the five days of treatment (Day 1 to Day 5) at bedtime
  Number, frequency and dosage of pain relief treatments assessed by patient diary
Assessment of satisfaction | through study completion (Day 6), an average of one week
  Assessment of satisfaction by Likert scale. It is a 7-point Likert scale (1: extremely dissatisfied, 2: very dissatisfied, 3: dissatisfied, 4: neutral, 5: satisfied, 6: very satisfied, 7: extremely satisfied).
Assessment of Clinical Global Impression of Improvement | through study completion (Day 6), an average of one week
  Assessment of Clinical Global Impression of Improvement by CGI scale. It is a 7-point scale (1=very much improved; 7=very much worse)
Incidence of adverse events and treatment adherence | during the five days of treatment (Day 1 to Day 5)
  Incidence of adverse events and treatment adherence collected by patients diary and phone

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Tivoli Ducos, Bordeaux, Gironde, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merlot B, Elie V, Perigord A, Husson Z, Jubert A, Chanavaz-Lacheray I, Dennis T, Cotty-Eslous M, Roman H. Pain Reduction With an Immersive Digital Therapeutic in Women Living With Endometriosis-Related Pelvic Pain: At-Home Self-Administered Randomized Controlled Trial. J Med Internet Res. 2023 Jun 28;25:e47869. doi: 10.2196/47869. PMID 37260160